CLINICAL TRIAL: NCT03492385
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of MEDI2452 (PB2452) With and Without Ticagrelor Pretreatment in Healthy Volunteers
Brief Title: Study to Evaluate the Safety, Tolerability, PK, and PD of PB2452 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SFJ Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PB2452-PT-CL-0001
Record Dates: First submitted 2018-04-02; First posted 2018-04-10 (Actual); Results first posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-08

CONDITIONS: Healthy
MeSH Terms: interventions — Aftercare

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- 1: 100 mg PB2452 or Placebo (no Ticagrelor) (Experimental): PB2452 Infusion or Placebo - Sodium Chloride
  Interventions: Drug: PB2452 Infusion; Drug: Placebo - Sodium Chloride
- 2: 300 mg PB2452 or Placebo (no Ticagrelor) (Experimental): PB2452 Infusion or Placebo - Sodium Chloride
  Interventions: Drug: PB2452 Infusion; Drug: Placebo - Sodium Chloride
- 3: 1000 mg PB2452 or Placebo (no Ticagrelor) (Experimental): PB2452 Infusion or Placebo - Sodium Chloride
  Interventions: Drug: PB2452 Infusion; Drug: Placebo - Sodium Chloride
- 4: 1000 mg PB2452 or Placebo (Ticagrelor Pre-Trx) (Experimental): PB2452 Infusion or Placebo - Sodium Chloride With Ticagrelor Oral Tablet: 180 mg+90 mg BID for a total of 5 doses
  Interventions: Drug: PB2452 Infusion; Drug: Placebo - Sodium Chloride
- 5: 3000 mg PB2452 or Placebo (Ticagrelor Pre-Trx) (Experimental): PB2452 Infusion or Placebo - Sodium Chloride with Ticagrelor Oral Tablet: 180 mg+90 mg BID for a total of 5 doses
  Interventions: Drug: PB2452 Infusion; Drug: Placebo - Sodium Chloride; Drug: Ticagrelor Oral Tablet - Pre-Treatment
- 6: 9000 mg PB2452 or Placebo (Ticagrelor Pre-Trx) (Experimental): PB2452 Infusion or Placebo - Sodium Chloride with Ticagrelor Oral Tablet: 180 mg+90 mg BID for a total of 5 doses
  Interventions: Drug: PB2452 Infusion; Drug: Placebo - Sodium Chloride; Drug: Ticagrelor Oral Tablet - Pre-Treatment
- 7: 18000 mg PB2452 or Placebo (Ticagrelor Pre-Trx) (Experimental): PB2452 Infusion or Placebo - Sodium Chloride with Ticagrelor Oral Tablet: 180 mg+90 mg BID for a total of 5 doses
  Interventions: Drug: PB2452 Infusion; Drug: Placebo - Sodium Chloride; Drug: Ticagrelor Oral Tablet - Pre-Treatment
- 8: Dose TBD mg PB2452 or Placebo (Ticagrelor Pre-Trx) (Experimental): PB2452 Infusion or Placebo - Sodium Chloride with Ticagrelor Oral Tablet: 180 mg+90 mg BID for 5 doses
  Interventions: Drug: PB2452 Infusion; Drug: Placebo - Sodium Chloride; Drug: Ticagrelor Oral Tablet - Pre-Treatment
- 9: Dose TBD mg PB2452 or Placebo (Ticagrelor Pre and Post-Trx) (Experimental): PB2452 Infusion or Placebo - Sodium Chloride with Ticagrelor Oral Tablet: 180 mg+90 mg BID for 5 doses and 180 mg 24 hours post-dose
  Interventions: Drug: PB2452 Infusion; Drug: Placebo - Sodium Chloride; Drug: Ticagrelor Oral Tablet - Pre-Treatment and Post-Treatment
- 10: Dose TBD mg PB2452 or Placebo (Ticagrelor Pre-Txt) (Experimental): PB2452 Infusion or Placebo - Sodium Chloride with Ticagrelor Oral Tablet: 180 mg+90 mg BID for 5 doses
  Interventions: Drug: PB2452 Infusion; Drug: Placebo - Sodium Chloride; Drug: Ticagrelor Oral Tablet - Pre-Treatment

INTERVENTIONS:
Drug: PB2452 Infusion — 30 minute - 12 hour infusion
Drug: Placebo - Sodium Chloride — 30 minute - 12 hour infusion
Drug: Ticagrelor Oral Tablet - Pre-Treatment — Ticagrelor 180 mg + 90 mg BID for 5 doses prior to MEDI2452 (PB2452) or Placebo
  Arms: 10: Dose TBD mg PB2452 or Placebo (Ticagrelor Pre-Txt); 5: 3000 mg PB2452 or Placebo (Ticagrelor Pre-Trx); 6: 9000 mg PB2452 or Placebo (Ticagrelor Pre-Trx); 7: 18000 mg PB2452 or Placebo (Ticagrelor Pre-Trx); 8: Dose TBD mg PB2452 or Placebo (Ticagrelor Pre-Trx)
Drug: Ticagrelor Oral Tablet - Pre-Treatment and Post-Treatment — Ticagrelor 180 mg + 90 mg BID for 5 doses prior to MEDI2452 (PB2452) or Placebo and Ticagerlor 180 mg 24 hours following MEDI2452 (PB2452) or Placebo
  Arms: 9: Dose TBD mg PB2452 or Placebo (Ticagrelor Pre and Post-Trx)

SUMMARY:
This is a Phase 1, first-in-human, randomized, double-blind, placebo-controlled, single ascending dose, sequential group study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of PB2452 with and without ticagrelor pretreatment when administered to healthy male and female subjects.

Up to 6 dose levels will be evaluated. This study will have up to 10 cohorts and up to a total of approximately 76 subjects with either 4 or 8 healthy young subjects in Cohorts 1 through 9 or approximately 16 older subjects in Cohort 10. The starting dose of PB2452 will be 100 mg and the planned doses for subsequent cohorts are 300, 1000, 3000, 9000, and 18000 mg.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is male or female between 18 and 50 years of age, inclusive.
2. The subject has a body mass index between 18 and 35 kg/m2 and a weight of ≥50 kg but ≤120 kg, inclusive, at screening.
3. The subject is considered by the investigator to be in good general health as determined by medical history, clinical laboratory test results, vital sign measurements, 12 lead ECG results, and physical examination findings at screening.

   Specific inclusionary laboratory values at screening and check-in require the following:
   * Aspartate transaminase (AST), alanine transaminase (ALT), total serum bilirubin and alkaline phosphatase levels within the normal range as defined by the clinical laboratory
   * White blood cell (WBC) count, platelet count and hemoglobin level within the normal range as defined by the clinical laboratory
   * Thyroid stimulating hormone (TSH) level within the normal range as defined by the clinical laboratory at screening
   * Prothrombin time (PT) and partial thromboplastin time (PTT) level within the normal range as defined by the clinical laboratory
4. Female subjects of childbearing potential must not be pregnant, lactating, or planning to become pregnant before 3 months after the last dose of study drug, and have a negative serum pregnancy test at screening and check-in. Female subjects of childbearing potential must use 2 effective methods of birth control (ie, oral, implantable, patch, or injectable contraceptives in combination with a condom, hormone-containing intrauterine device that has been in place for at least 2 months prior to screening in combination with a condom, double-barrier method [ie, condoms, sponge, diaphragm, or cervical cap with spermicidal gels or cream], or vasectomy for male subjects or male partners of female subjects) from 30 days before study drug administration through the end of the study. Women are considered not to be of childbearing potential if they have fulfilled one of the following criteria: documentation of irreversible surgical sterilization (ie, hysterectomy, or bilateral oophorectomy [not tubal ligation]), or postmenopausal (defined as amenorrhea for 12 consecutive months following cessation of all exogenous hormonal treatments, and documented plasma follicle-stimulating hormone level >40 IU/mL or amenorrhea for 24 consecutive months). Male subjects with partners of childbearing potential must agree to use appropriate and effective measures of contraception (eg, condom plus diaphragm with spermicide; condom plus spermicide) during the study and for 30 days after the last dose of study drug, and to refrain from donating sperm for at least 7 days prior to the first dose of study drug until at least 90 days following the last dose of study drug.
5. The subject agrees to comply with all protocol requirements.
6. The subject is able to provide written informed consent.

Exclusion Criteria:

1. History of any clinically significant acute or chronic disease or medical disorder.
2. History or presence of gastrointestinal, hepatic (with the exception of Gilbert's syndrome), or renal disease or renal insufficiency (ie, estimated glomerular filtration rate <60 ml/min/1.73m2), or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
3. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of study drug or any planned surgical procedure that will occur during the study (from screening through the Day 28 follow up visit).
4. Any clinically significant abnormal findings in physical examination, vital signs, laboratory assessments, and ECG parameters identified during screening or check-in.
5. Any history of arterial or venous thrombosis, including any of the following:

   * History of transient ischemic attack, cardiovascular accident, stroke (ischemic or hemorrhagic), unstable angina, myocardial infarction, or peripheral arterial disease
   * History of deep venous thrombosis, pulmonary embolus, thrombophlebitis, or cavernous malformations
6. Any increased risk of bleeding, including the following:

   * Recent history (within 30 days preceding the first dose of study drug) of gastrointestinal bleeding
   * Any history of severe head trauma, intracranial hemorrhage, intracranial neoplasm, arteriovenous malformation, aneurysm, or proliferative retinopathy
   * Any history of intracranial, intraocular, retroperitoneal, or spinal bleeding
   * Any recent (within 30 days preceding the first dose of study drug) major trauma
   * History of hemorrhagic disorders that may increase the risk of bleeding (eg, hemophilia, von Willebrand's disease)
   * Receiving chronic treatment with nonsteroidal anti-inflammatory drugs (including aspirin [greater than 100 mg daily]), anticoagulants, or other antiplatelet agents that cannot be discontinued (including clopidogrel, prasugrel, ticlopidine, dipyridamole, or cilostazol).
   * Have taken, within 30 days of screening, any oral or parenteral anticoagulant, including low molecular-weight heparin
   * Have taken non-steroidal anti-inflammatory medications, including aspirin, within 14 days of screening
7. The subject has a positive test result for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus types 1 or 2 antibodies at screening.
8. Any ongoing or recent (ie, during the screening period) minor medical complaints that may interfere with the interpretation of the study data or are considered unlikely to comply with study procedures, restrictions, and requirements as judged by the investigator.
9. Concomitant oral or IV therapy with strong CYP3A inhibitors, CYP3A substrates with narrow therapeutic indices, or strong CYP3A inducers, which cannot be stopped within at least 5 half-lives, but not shorter than 10 days, before randomization (a list of examples can be found in Section 6.2).
10. Any prescription (excluding hormonal birth control) or over the counter medications (except paracetamol [up to 2 g per day]), including herbal or nutritional supplements, within 14 days before the first dose of study drug.
11. The subject has consumed grapefruit or grapefruit juice, Seville orange or Seville orange containing products (eg, marmalade), or alcohol-, or xanthine containing products within 48 hours before dosing with study drug.
12. The subject is participating in any other study or is taking part in a non medication study which, in the opinion of the investigator, would interfere with the outcome of the study.
13. The subject has received another new chemical entity (defined as a compound which has not been approved for marketing) or any marketed or investigational biologic agent within 30 days of the first administration of study drug in this study. The period of exclusion begins 30 days after the final dose or 5 half-lives of the experimental medication has elapsed, whichever is longer.
14. The subject has involvement with any PhaseBio or study site employee or their close relatives (eg, spouse, parents, siblings, or children whether biological or legally adopted).
15. The subject has previously received MEDI2452 (PB2452).
16. The subject is a smoker or has used nicotine or nicotine containing products (eg, snuff, nicotine patch, nicotine chewing gum, mock cigarettes, or inhalers) within 3 months before the first dose of study drug.
17. The subject has a known or suspected history of drug abuse (including alcohol) or has a positive test result for drugs of abuse, alcohol, or cotinine (nicotine level above 300 ng/mL) at screening or check-in.
18. The subject has been involved in strenuous activity or contact sports within 24 hours before the first dose of study drug and while confined in the clinical site.
19. The subject has donated blood or plasma within 1 month of screening or any blood donation/loss more than 500 mL during the 3 months prior to the first dose of study drug.
20. The subject has a history of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the investigator or history of hypersensitivity to drugs with a similar chemical structure or class to ticagrelor, any biologic therapeutic agent, or any significant food allergy that could preclude a standard diet in the clinical site.
21. Concern for the inability of the subject to comply with study procedures and/or follow up, or, in the opinion of the investigator, the subject is not suitable for entry into the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 64 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2018-09-18 (Actual); Study Completion 2018-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: LuAnn Bundrant, MD, Principal Investigator — PPD Development, LP
Locations (1):
- PPD, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bhatt DL, Pollack CV, Weitz JI, Jennings LK, Xu S, Arnold SE, Umstead BR, Mays MC, Lee JS. Antibody-Based Ticagrelor Reversal Agent in Healthy Volunteers. N Engl J Med. 2019 May 9;380(19):1825-1833. doi: 10.1056/NEJMoa1901778. Epub 2019 Mar 17. PMID 30883047

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Healthy participants who met all the inclusion criteria and none of the exclusion criteria were randomly assigned to receive either PB2452 or placebo in a ratio of 3:1 in all treatment cohorts.
Groups:
- Cohort 1: 100 mg PB2452 (no Ticagrelor): PB2452 Infusion: single 30-minute intravenous (IV) infusion of 100 mg PB2452
- Cohort 2: 300 mg PB2452 (no Ticagrelor): PB2452 Infusion: single 30-minute IV infusion of 300 mg PB2452
- Cohort 3: 1000 mg PB2452 (no Ticagrelor): PB2452 Infusion: single 30-minute IV infusion of 1000 mg PB2452
- Cohort 1 to 3: Placebo; Cohort 4 to 6: Placebo: Placebo - Sodium Chloride: single 30-minute IV infusion of placebo
- Cohort 4: 1000 mg PB2452 (Ticagrelor Pre-Trx): PB2452 Infusion: single 30-minute IV infusion of 1000 mg PB2452
  Ticagrelor Oral Tablet - Pre-Treatment: Ticagrelor 180 mg + 90 mg twice daily (BID) for 5 doses prior to administration of a single IV dose of PB2452
- Cohort 5: 3000 mg PB2452 (Ticagrelor Pre-Trx): PB2452 Infusion: single 30-minute IV infusion of 3000 mg PB2452
  Ticagrelor Oral Tablet - Pre-Treatment: Ticagrelor 180 mg + 90 mg BID for 5 doses prior to administration of a single IV dose of PB2452
- Cohort 6: 9000 mg PB2452 (Ticagrelor Pre-Trx): PB2452 Infusion: single 30-minute IV infusion of 9000 mg PB2452
  Ticagrelor Oral Tablet - Pre-Treatment: Ticagrelor 180 mg + 90 mg BID for 5 doses prior to administration of a single IV dose of PB2452
- Cohort 7: 18000 mg PB2452 (Ticagrelor Pre-Trx): PB2452 Infusion: single IV infusion of 18000 mg PB2452 for 8 hours
  Ticagrelor Oral Tablet - Pre-Treatment: Ticagrelor 180 mg + 90 mg BID for 5 doses prior to administration of a single IV dose of PB2452
- Cohort 8: 18000 mg PB2452 (Ticagrelor Pre-Trx): PB2452 Infusion: single IV infusion of 18000 mg PB2452 for 12 hours
  Ticagrelor Oral Tablet - Pre-Treatment: Ticagrelor 180 mg + 90 mg BID for 5 doses prior to administration of a single IV dose of PB2452
- Cohort 9: 18000 mg PB2452 (Ticagrelor Pre-Trx): PB2452 Infusion: single IV infusion of 18000 mg PB2452 for 16 hours and 20 minutes
  Ticagrelor Oral Tablet - Pre-Treatment: Ticagrelor 180 mg + 90 mg BID for 5 doses prior to administration of a single IV dose of PB2452
- Cohort 10: 18000 mg PB2452 (Ticagrelor Pre-Trx): PB2452 Infusion: single IV infusion of 18000 mg PB2452 for 16 hours and 12 minutes
  Ticagrelor Oral Tablet - Pre-Treatment: Ticagrelor 180 mg + 90 mg BID for 5 doses prior to administration of a single IV dose of PB2452
- Cohort 7 to 10: Placebo: Placebo - Sodium Chloride: single 8-hour to 16.5-hour IV infusion of placebo
Period: Overall Study
Arm/Group | Cohort 1: 100 mg PB2452 (no Ticagrelor) | Cohort 2: 300 mg PB2452 (no Ticagrelor) | Cohort 3: 1000 mg PB2452 (no Ticagrelor) | Cohort 1 to 3: Placebo | Cohort 4: 1000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 5: 3000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 6: 9000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 4 to 6: Placebo | Cohort 7: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 8: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 9: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 10: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 7 to 10: Placebo
Started | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 3 | 6 | 7
Completed | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 3 | 6 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population: all participants who received any amount of study drug.
Groups:
- Cohort 1: 100 mg PB2452 (no Ticagrelor): PB2452 Infusion: single 30-minute IV infusion of 100 mg PB2452
- Cohort 4: 1000 mg PB2452 (Ticagrelor Pre-Trx): PB2452 Infusion: single 30-minute IV infusion of 1000 mg PB2452
  Ticagrelor Oral Tablet - Pre-Treatment: Ticagrelor 180 mg + 90 mg BID for 5 doses prior to administration of a single IV dose of PB2452
- Total: Total of all reporting groups
Arm/Group | Cohort 1: 100 mg PB2452 (no Ticagrelor) | Cohort 2: 300 mg PB2452 (no Ticagrelor) | Cohort 3: 1000 mg PB2452 (no Ticagrelor) | Cohort 1 to 3: Placebo | Cohort 4: 1000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 5: 3000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 6: 9000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 4 to 6: Placebo | Cohort 7: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 8: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 9: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 10: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 7 to 10: Placebo | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 3 | 6 | 7 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.7 (2.89) | 30.0 (10.58) | 40.0 (12.49) | 28.0 (9.17) | 30.7 (5.99) | 30.2 (9.95) | 33.8 (11.96) | 30.7 (5.79) | 26.7 (8.87) | 29.7 (8.04) | 30.7 (5.86) | 28.7 (9.03) | 39.4 (7.16) | 31.4 (8.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 1 | 3 | 3 | 5 | 2 | 2 | 3 | 2 | 2 | 2 | 30
  Male | 2 | 1 | 1 | 2 | 3 | 3 | 1 | 4 | 4 | 3 | 1 | 4 | 5 | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population of participants based on their ethnicity.
  Participants
    Hispanic or Latino | 2 | 1 | 2 | 1 | 3 | 3 | 4 | 2 | 2 | 2 | 2 | 1 | 3 | 28
    Not Hispanic or Latino | 1 | 2 | 1 | 2 | 3 | 3 | 2 | 4 | 4 | 4 | 1 | 5 | 4 | 36
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population of participants based on their race.
  Participants
    White | 1 | 2 | 2 | 1 | 4 | 3 | 5 | 4 | 3 | 1 | 3 | 3 | 2 | 34
    Black or African American | 2 | 1 | 1 | 2 | 2 | 2 | 0 | 1 | 3 | 4 | 0 | 3 | 5 | 26
    Asian | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    Multiple | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug-related.
Time Frame: Day -3 (Cohorts 4 through 10) or Day -1 (Cohorts 1 through 3) until Day 28
Population: Safety population: all participants who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: 100 mg PB2452 (no Ticagrelor) | Cohort 2: 300 mg PB2452 (no Ticagrelor) | Cohort 3: 1000 mg PB2452 (no Ticagrelor) | Cohort 1 to 3: Placebo | Cohort 4: 1000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 5: 3000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 6: 9000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 4 to 6: Placebo | Cohort 7: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 8: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 9: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 10: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 7 to 10: Placebo
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 3 | 6 | 7
Participants
  Any Treatment-Emergent AE | 0 | 0 | 1 | 1 | 3 | 0 | 6 | 1 | 2 | 2 | 1 | 2 | 0
  Any study-drug-related TEAE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any severe TEAE | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any SAE | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any AE leading to early study discontinuation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any dose limiting toxicity | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities
Description: Number of participants with clinically significant abnormal laboratory findings for hematology, coagulation, serum chemistry, urinalysis and drug tests.
Time Frame: 30 Day - Starting day of dosing
Population: Safety population: all participants who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: 100 mg PB2452 (no Ticagrelor) | Cohort 2: 300 mg PB2452 (no Ticagrelor) | Cohort 3: 1000 mg PB2452 (no Ticagrelor) | Cohort 1 to 3: Placebo | Cohort 4: 1000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 5: 3000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 6: 9000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 4 to 6: Placebo | Cohort 7: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 8: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 9: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 10: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 7 to 10: Placebo
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 3 | 6 | 7
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Change in Diastolic Blood Pressure
Description: Diastolic blood pressure measurements were measured at specific time points.
Time Frame: Days 1, 2, 3, 4, 7 and 28
Population: Safety population: all participants who received any amount of study drug.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Cohort 1: 100 mg PB2452 (no Ticagrelor) | Cohort 2: 300 mg PB2452 (no Ticagrelor) | Cohort 3: 1000 mg PB2452 (no Ticagrelor) | Cohort 1 to 3: Placebo | Cohort 4: 1000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 5: 3000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 6: 9000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 4 to 6: Placebo | Cohort 7: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 8: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 9: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 10: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 7 to 10: Placebo
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 3 | 6 | 7
mmHg
  Change from Baseline - Day 1/0.5 Hour: number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6 | 4 | 4 | 3 | 6 | 7
  Change from Baseline - Day 1/0.5 Hour | 1.7 (6.66) | -2.3 (7.57) | 5.7 (3.21) | -1.7 (10.02) | -0.8 (7.76) | -2.7 (5.39) | -0.5 (3.39) | -1.3 (5.13) | -2.5 (3.70) | 4.5 (3.51) | -4.0 (4.58) | -2.5 (5.96) | -1.4 (8.30)
  Change from Baseline - Day 1/0.75 Hour | 0.7 (10.21) | -1.0 (8.89) | 3.3 (6.43) | -0.3 (9.07) | 0.3 (9.29) | -1.0 (1.79) | -1.2 (3.54) | 1.3 (5.54) | 1.5 (9.97) | -0.3 (7.28) | -2.3 (1.53) | -2.0 (6.48) | -0.4 (8.92)
  Change from Baseline - Day 1/1 Hour | -0.7 (11.37) | 0 (4.58) | 2.7 (6.66) | 4.0 (6.24) | 3.5 (8.78) | 0.3 (3.33) | 0.3 (3.98) | 2.8 (6.43) | 3.8 (11.18) | 0.5 (5.54) | -6.7 (1.53) | -1.7 (6.83) | 2.1 (9.69)
  Change from Baseline - Day 1/2 Hour: number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 3 | 5 | 7
  Change from Baseline - Day 1/2 Hour | 12.7 (7.23) | 1.0 (2.00) | 0.7 (1.53) | -1.7 (8.14) | 1.0 (6.84) | -1.5 (3.94) | 0 (3.58) | -0.3 (3.33) | 2.7 (9.58) | -1.0 (6.54) | -5.3 (1.53) | -2.6 (4.67) | 2.9 (9.39)
  Change from Baseline - Day 1/4 Hour | 1.3 (3.21) | -9.0 (2.00) | -0.3 (1.53) | -3.3 (8.02) | -2.2 (5.53) | -3.3 (4.72) | -0.5 (5.47) | -1.5 (4.04) | -3.8 (7.31) | -1.5 (6.16) | -8.7 (5.51) | 1.3 (9.69) | 0.7 (9.60)
  Change from Baseline - Day 1/8 Hour: number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 5 | 3 | 6 | 7
  Change from Baseline - Day 1/8 Hour | 0.3 (7.02) | -8.7 (4.93) | -1.3 (4.51) | 2.7 (4.62) | -4.2 (9.91) | -3.3 (8.02) | -0.2 (5.67) | -0.7 (6.02) | -3.7 (6.02) | -3.2 (5.72) | -10.3 (5.03) | -3.2 (5.60) | -3.1 (12.19)
  Change from Baseline - Day 2/24 Hour | 3.0 (5.57) | -2.7 (4.73) | 2.3 (1.15) | -2.7 (4.04) | 1.2 (5.08) | -2.3 (4.37) | -0.3 (5.28) | 1.7 (6.12) | -2.2 (3.31) | -2.3 (8.14) | -3.3 (6.66) | -3.3 (5.57) | -1.7 (8.75)
  Change from Baseline - Day 2/30 Hour | 4.0 (4.36) | -5.7 (8.02) | -4.7 (4.04) | -6.7 (9.61) | -2.2 (5.60) | -4.5 (6.22) | -2.5 (4.93) | -5.3 (4.68) | -6.2 (2.56) | -5.0 (8.58) | -7.7 (8.74) | -3.0 (4.98) | -3.1 (13.04)
  Change from Baseline - Day 2/36 Hour | 3.3 (5.51) | -7.7 (5.86) | -0.7 (5.03) | -5.3 (6.81) | 0.2 (9.06) | -2.0 (5.66) | -3.5 (5.13) | -4.3 (7.03) | -4.3 (4.13) | -7.0 (7.13) | -11.7 (8.08) | -5.8 (3.66) | -4.7 (8.20)
  Change from Baseline - Day 3/42 Hour | 1.0 (12.12) | -9.3 (1.53) | -6.0 (3.46) | -3.3 (7.02) | -7.2 (7.81) | -3.2 (3.87) | -1.2 (5.95) | -5.5 (3.45) | -4.0 (4.43) | -6.2 (10.96) | -12.7 (3.21) | -8.0 (10.20) | -9.7 (8.90)
  Change from Baseline - Day 3/48 Hour | 5.0 (5.29) | -1.0 (4.00) | -1.7 (6.43) | -3.3 (13.50) | 3.8 (7.14) | -0.2 (4.83) | 5.8 (10.01) | -0.2 (3.97) | -1.8 (3.97) | -0.2 (4.71) | -7.0 (3.46) | -4.5 (6.41) | -2.3 (9.79)
  Change from Baseline - Day 4 | 7.7 (9.45) | 3.7 (4.16) | 2.7 (3.06) | 5.3 (3.79) | 8.2 (5.42) | 5.8 (5.71) | 4.7 (4.97) | 2.0 (6.16) | 3.8 (4.40) | -4.2 (7.78) | -10.3 (4.16) | -0.8 (6.40) | -1.9 (9.62)
  Change from Baseline - Day 7: number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6 | 5 | 6 | 3 | 6 | 7
  Change from Baseline - Day 7 | 9.0 (10.58) | -1.3 (6.81) | 6.3 (3.06) | 6.0 (6.08) | 7.0 (5.44) | 3.2 (7.08) | 4.2 (3.87) | 0.7 (7.34) | 0.2 (7.33) | 6.5 (8.57) | -5.0 (15.62) | 5.3 (10.63) | 7.4 (14.39)
  Change from Baseline - Day 28 | 12.0 (7.94) | 5.0 (2.65) | 1.3 (1.53) | 4.0 (4.58) | 8.8 (7.08) | 6.7 (5.61) | 4.7 (5.43) | 5.7 (4.89) | 3.5 (3.83) | 7.8 (5.98) | -5.0 (12.00) | 9.2 (6.85) | 4.9 (10.17)

4. Primary Outcome: Change in Systolic Blood Pressure
Description: Systolic blood pressure measurements were measured at specific time points.
Time Frame: Days 1, 2, 3, 4, 7 and 28
Population: Safety population: all participants who received any amount of study drug.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Cohort 1: 100 mg PB2452 (no Ticagrelor) | Cohort 2: 300 mg PB2452 (no Ticagrelor) | Cohort 3: 1000 mg PB2452 (no Ticagrelor) | Cohort 1 to 3: Placebo | Cohort 4: 1000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 5: 3000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 6: 9000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 4 to 6: Placebo | Cohort 7: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 8: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 9: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 10: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 7 to 10: Placebo
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 3 | 6 | 7
mmHg
  Change from Baseline - Day 1/0.5 Hour: number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6 | 4 | 4 | 3 | 6 | 7
  Change from Baseline - Day 1/0.5 Hour | 3.0 (15.10) | -0.7 (8.33) | 6.7 (6.51) | 0.3 (12.86) | -4.8 (4.75) | -0.3 (2.42) | 1.3 (2.73) | -3.0 (6.87) | 1.5 (6.61) | -0.3 (8.30) | 4.7 (7.37) | -1.7 (4.63) | -0.7 (4.68)
  Change from Baseline - Day 1/0.75 Hour | 4.0 (5.00) | 2.0 (4.36) | 2.3 (6.03) | 1.0 (13.23) | -1.2 (6.24) | 0.2 (3.43) | 2.8 (2.93) | 1.3 (8.12) | 11.5 (12.93) | -1.2 (11.13) | -6.0 (5.29) | -3.3 (4.80) | -1.4 (7.28)
  Change from Baseline - Day 1/1 Hour | 7.7 (5.13) | 2.7 (3.06) | 3.0 (4.58) | 2.0 (4.36) | 2.7 (5.20) | 1.7 (5.61) | 1.2 (1.72) | -0.5 (6.44) | 8.0 (12.21) | 0.2 (6.85) | 4.7 (7.57) | -1.7 (6.65) | 1.0 (9.04)
  Change from Baseline - Day 1/2 Hour: number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 3 | 5 | 7
  Change from Baseline - Day 1/2 Hour | 5.7 (10.21) | -1.3 (4.93) | 1.7 (9.07) | -0.3 (5.86) | -2.5 (10.19) | -1.2 (4.45) | 0.3 (5.79) | -1.7 (5.61) | 7.8 (7.44) | -3.2 (10.15) | -4.7 (2.52) | 1.0 (2.12) | 1.0 (6.22)
  Change from Baseline - Day 1/4 Hour | 5.7 (9.87) | -4.0 (3.61) | 1.3 (3.21) | -1.3 (8.14) | -2.3 (3.50) | -1.5 (4.32) | -1.3 (5.13) | -0.8 (7.78) | 0.3 (3.14) | -1.7 (13.29) | -7.0 (16.52) | 1.2 (6.49) | 0.1 (11.35)
  Change from Baseline - Day 1/8 Hour: number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 5 | 3 | 6 | 7
  Change from Baseline - Day 1/8 Hour | 0.7 (11.02) | -1.0 (4.36) | -2.0 (1.73) | -1.3 (18.77) | -2.2 (11.05) | -2.3 (3.67) | 1.8 (10.30) | 0 (6.32) | -0.8 (6.18) | -4.8 (10.28) | -11.7 (8.62) | 0.8 (6.62) | -0.7 (11.43)
  Change from Baseline - Day 2/24 Hour | 4.7 (5.13) | -3.7 (11.59) | 5.7 (7.77) | 3.7 (9.61) | -2.8 (3.71) | -1.7 (5.96) | 3.5 (8.46) | 1.8 (8.35) | 1.3 (6.09) | -7.0 (16.46) | 1.7 (12.86) | -0.5 (8.60) | 1.9 (7.95)
  Change from Baseline - Day 2/30 Hour | 4.0 (12.12) | 1.0 (10.15) | 0.7 (4.51) | 4.3 (12.10) | -3.3 (6.86) | -4.2 (11.27) | -0.7 (6.22) | -4.0 (8.79) | -1.5 (2.26) | -3.7 (13.91) | -0.7 (15.95) | -4.0 (6.13) | -3.3 (14.07)
  Change from Baseline - Day 2/36 Hour | 1.0 (6.08) | -0.7 (7.77) | 5.0 (6.00) | -2.7 (5.86) | 3.8 (10.40) | 2.2 (5.23) | -2.8 (8.52) | -0.2 (11.62) | 1.0 (4.10) | -3.0 (11.26) | -0.7 (15.14) | 1.5 (9.97) | 1.9 (13.12)
  Change from Baseline - Day 3/42 Hour | 2.3 (9.07) | -9.7 (2.52) | 3.0 (12.12) | -6.0 (4.58) | -8.2 (8.77) | -3.3 (8.31) | -3.0 (6.69) | -3.8 (10.46) | -7.7 (7.63) | -10.0 (12.96) | -2.7 (14.15) | -7.3 (14.79) | -7.7 (17.97)
  Change from Baseline - Day 3/48 Hour | 2.0 (8.72) | 5.3 (7.57) | 0.3 (7.77) | 0.3 (3.21) | 3.8 (7.78) | 3.7 (7.97) | 4.3 (8.98) | 1.5 (6.25) | 1.0 (5.90) | -0.5 (11.26) | 3.0 (11.53) | -2.3 (12.42) | -1.1 (12.39)
  Change from Baseline - Day 4 | 15.0 (2.65) | 1.0 (5.57) | 2.3 (9.07) | 6.3 (3.79) | 1.0 (3.95) | 2.3 (5.16) | -2.3 (6.98) | 6.7 (11.34) | 2.7 (10.58) | -5.3 (11.22) | -4.3 (14.47) | 1.3 (7.87) | -4.4 (12.95)
  Change from Baseline - Day 7: number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6 | 5 | 6 | 3 | 6 | 7
  Change from Baseline - Day 7 | 11.7 (5.51) | 5.7 (15.50) | 6.3 (13.50) | 7.7 (7.51) | 4.8 (5.91) | 5.2 (6.68) | 0.2 (4.58) | 1.7 (10.97) | 1.6 (10.21) | 3.5 (12.82) | 3.3 (16.62) | 4.5 (8.69) | 10.1 (13.80)
  Change from Baseline - Day 28 | 12.0 (7.21) | 6.3 (6.51) | 1.0 (8.19) | 0.7 (8.74) | 10.0 (10.55) | 3.5 (9.83) | 6.0 (7.46) | 0.8 (8.38) | 8.7 (4.93) | 3.8 (10.19) | -0.3 (17.01) | 8.7 (11.04) | 10.6 (12.91)

5. Primary Outcome: Change In Oral Body Temperature
Description: Body temperature measurements were measured at specific time points.
Time Frame: Days 1, 2, 3, 4, 7 and 28
Population: Safety population: all participants who received any amount of study drug.
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Cohort 1: 100 mg PB2452 (no Ticagrelor) | Cohort 2: 300 mg PB2452 (no Ticagrelor) | Cohort 3: 1000 mg PB2452 (no Ticagrelor) | Cohort 1 to 3: Placebo | Cohort 4: 1000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 5: 3000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 6: 9000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 4 to 6: Placebo | Cohort 7: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 8: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 9: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 10: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 7 to 10: Placebo
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 3 | 6 | 7
Degrees Celsius
  Change from Baseline - Day 1/0.5 Hour: number analyzed (Participants) | 0 | 0 | 3 | 1 | 6 | 6 | 6 | 6 | 4 | 4 | 3 | 6 | 7
  Change from Baseline - Day 1/0.5 Hour |  |  | -0.23 (0.321) | 0.30 (NA) — The "n" for this parameter at Day 1/0.5h is 1, therefore, there is no standard deviation. | 0.12 (0.183) | -0.05 (0.217) | -0.15 (0.207) | -0.02 (0.313) | 0.05 (0.265) | -0.03 (0.465) | -0.17 (0.473) | -0.10 (0.141) | -0.41 (1.512)
  Change from Baseline - Day 1/0.75 Hour | 0.03 (0.231) | -0.20 (0.361) | 0.13 (0.115) | 0 (0.265) | 0.12 (0.248) | 0.07 (0.234) | -0.03 (0.301) | 0.03 (0.273) | 0.07 (0.186) | 0.03 (0.242) | 0.10 (0.173) | 0.03 (0.186) | 0.03 (0.304)
  Change from Baseline - Day 1/1 Hour | -0.13 (0.306) | -0.17 (0.208) | 0.07 (0.231) | -0.57 (1.002) | 0.07 (0.186) | -0.05 (0.308) | -0.13 (0.121) | 0 (0.434) | 0 (0.228) | -0.07 (0.197) | 0.10 (0.265) | -0.05 (0.207) | 0.01 (0.402)
  Change from Baseline - Day 1/2 Hour: number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 3 | 5 | 7
  Change from Baseline - Day 1/2 Hour | -0.03 (0.379) | -0.03 (0.115) | 0.17 (0.351) | 0.10 (0) | 0.05 (0.187) | -0.02 (0.248) | -0.03 (0.207) | 0.10 (0.341) | 0.07 (0.339) | -0.08 (0.194) | 0.10 (0.200) | -0.20 (0.274) | 0 (0.277)
  Change from Baseline - Day 1/4 Hour | 0.17 (0.289) | -0.20 (0.200) | 0.07 (0.058) | 0.17 (0.153) | 0.10 (0.155) | 0.18 (0.271) | 0.07 (0.294) | 0.20 (0.253) | 0.07 (0.403) | 0.22 (0.479) | 0.20 (0.361) | 0.13 (0.361) | 0.13 (0.350)
  Change from Baseline - Day 1/8 Hour: number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 5 | 3 | 6 | 7
  Change from Baseline - Day 1/8 Hour | 0.30 (0.436) | 0.07 (0.153) | 0.03 (0.153) | 0.60 (0.624) | 0.18 (0.248) | 0.33 (0.585) | -0.07 (0.383) | -0.07 (0.225) | 0.17 (0.273) | 0.04 (0.288) | 0.27 (0.058) | 0.03 (0.288) | 0.10 (0.346)
  Change from Baseline - Day 2/24 Hour | -0.13 (0.306) | -0.43 (0.058) | -0.13 (0.306) | -0.17 (0.404) | 0.20 (0.297) | -0.08 (0.264) | -0.18 (0.325) | -0.15 (0.226) | -0.32 (0.397) | -0.15 (0.356) | -0.10 (0.100) | -0.18 (0.454) | -0.30 (0.416)
  Change from Baseline - Day 2/30 Hour | 0.30 (0.608) | -0.30 (0.100) | -0.17 (0.058) | 0.27 (0.153) | 0.30 (0.303) | 0.20 (0.316) | -0.17 (0.592) | -0.03 (0.361) | 0.02 (0.343) | 0 (0.590) | -0.17 (0.404) | -0.15 (0.251) | -0.07 (0.419)
  Change from Baseline - Day 2/36 Hour | 0.17 (0.666) | -0.47 (0.351) | 0.30 (0.361) | 0.23 (0.306) | 0.18 (0.232) | 0.03 (0.280) | -0.10 (0.253) | 0.07 (0.273) | -0.10 (0.283) | -0.27 (0.250) | 0.13 (0.416) | -0.03 (0.423) | -0.11 (0.463)
  Change from Baseline - Day 3/42 Hour | -0.10 (0.400) | -0.83 (0.231) | -0.30 (0.200) | -0.33 (0.603) | -0.37 (0.314) | -0.23 (0.333) | -0.43 (0.403) | -0.38 (0.343) | -0.57 (0.163) | -0.28 (0.454) | -0.37 (0.208) | -0.52 (0.232) | -0.29 (0.353)
  Change from Baseline - Day 3/48 Hour | -0.20 (0.529) | -0.27 (0.058) | -0.13 (0.208) | -0.20 (0.200) | 0.18 (0.172) | -0.20 (0.261) | -0.37 (0.497) | -0.10 (0.374) | 0.03 (0.333) | -0.20 (0.276) | 0.10 (0.100) | -0.23 (0.372) | -0.01 (0.344)
  Change from Baseline - Day 4 | 0 (0.300) | -0.27 (0.153) | 0.07 (0.404) | -0.27 (0.651) | 0.10 (0.438) | 0.08 (0.417) | -0.15 (0.327) | -0.12 (0.488) | -0.33 (0.294) | -0.08 (0.293) | 0.33 (0.306) | -0.20 (0.283) | 0.03 (0.293)
  Change from Baseline - Day 7: number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6 | 5 | 6 | 3 | 6 | 7
  Change from Baseline - Day 7 | -0.03 (0.551) | -0.53 (0.404) | 0 (0.265) | -0.50 (0.700) | -0.13 (0.333) | 0.50 (0.363) | -0.32 (0.293) | -0.08 (0.147) | -0.04 (0.241) | -0.33 (0.367) | 0.37 (0.231) | -0.43 (0.468) | -0.14 (0.294)
  Change from Baseline - Day 28 | -0.20 (0.624) | -0.43 (0.058) | -0.10 (0.200) | -0.37 (0.569) | -0.20 (0.303) | 0.03 (0.408) | -0.03 (0.383) | -0.18 (0.293) | -0.08 (0.458) | -0.45 (0.302) | -0.07 (0.651) | -0.35 (0.509) | -0.13 (0.390)

6. Primary Outcome: Change In Respiratory Rate
Description: Respiratory rate measurements were measured at specific time points.
Time Frame: Days 1, 2, 3, 4, 7 and 28
Population: Safety population: all participants who received any amount of study drug.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Cohort 1: 100 mg PB2452 (no Ticagrelor) | Cohort 2: 300 mg PB2452 (no Ticagrelor) | Cohort 3: 1000 mg PB2452 (no Ticagrelor) | Cohort 1 to 3: Placebo | Cohort 4: 1000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 5: 3000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 6: 9000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 4 to 6: Placebo | Cohort 7: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 8: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 9: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 10: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 7 to 10: Placebo
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 3 | 6 | 7
Breaths per minute
  Change from Baseline - Day 1/0.5 Hour: number analyzed (Participants) | 3 | 3 | 3 | 1 | 6 | 6 | 6 | 6 | 4 | 4 | 3 | 6 | 7
  Change from Baseline - Day 1/0.5 Hour | 0 (0) | 0 (0) | -2.0 (0) | -2.0 (NA) — The "n" for this parameter at Day 1/0.5h is 1, therefore, there is no standard deviation. | -1.3 (3.27) | 0.3 (2.94) | 0 (0) | -1.0 (2.10) | 0.5 (1.91) | -1.0 (1.15) | -0.7 (3.06) | -0.7 (3.01) | -0.6 (3.60)
  Change from Baseline - Day 1/0.75 Hour | -0.7 (2.31) | 3.3 (1.15) | -1.3 (3.06) | -1.3 (4.16) | -1.3 (4.32) | 0 (2.19) | 0.7 (1.63) | -1.7 (2.94) | -0.7 (3.50) | -1.0 (2.45) | -2.0 (4.00) | -0.3 (3.20) | -0.9 (2.27)
  Change from Baseline - Day 1/1 Hour | -3.3 (2.31) | 2.7 (2.31) | 0.7 (3.06) | -1.3 (4.16) | -1.0 (3.95) | 0.3 (2.34) | 1.3 (1.03) | -0.3 (2.94) | -0.7 (2.07) | 0 (2.83) | -2.7 (3.06) | -1.0 (3.29) | 0.3 (3.90)
  Change from Baseline - Day 1/2 Hour: number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 3 | 5 | 7
  Change from Baseline - Day 1/2 Hour | -1.3 (1.15) | 0 (2.00) | 0.7 (2.31) | 0 (2.00) | -1.3 (3.01) | 1.3 (3.27) | 3.3 (1.63) | 0 (3.35) | 0.7 (3.01) | 0.3 (2.66) | -0.7 (5.03) | -0.8 (3.03) | 1.4 (3.60)
  Change from Baseline - Day 1/4 Hour | -0.7 (1.15) | 0 (2.00) | -2.0 (2.00) | -0.7 (3.06) | -2.3 (4.63) | 1.0 (2.10) | 1.7 (2.34) | 0 (1.26) | 0.3 (4.27) | 0.3 (0.82) | 2.0 (4.00) | -2.3 (2.34) | -0.3 (3.73)
  Change from Baseline - Day 1/8 Hour: number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 5 | 3 | 6 | 7
  Change from Baseline - Day 1/8 Hour | 1.3 (3.06) | 5.3 (1.15) | -2.0 (4.00) | 1.3 (7.02) | -0.3 (2.94) | 3.0 (2.76) | -1.0 (2.76) | 0.3 (3.20) | 2.0 (2.53) | -2.0 (5.83) | -2.0 (5.29) | -0.3 (0.82) | 0.6 (4.58)
  Change from Baseline - Day 2/24 Hour | -2.0 (0) | 1.3 (3.06) | -0.7 (2.31) | 0.7 (2.31) | -3.0 (3.03) | -1.0 (2.10) | 2.3 (2.66) | -1.0 (2.10) | -1.0 (2.10) | -1.0 (3.03) | -3.3 (1.15) | -1.3 (4.32) | -1.4 (2.51)
  Change from Baseline - Day 2/30 Hour | 2.7 (3.06) | 3.3 (2.31) | 0.7 (1.15) | 1.3 (5.03) | 0.7 (4.84) | 1.0 (2.10) | 2.7 (2.42) | 0 (5.51) | -2.7 (2.73) | 1.7 (2.34) | -0.7 (4.62) | 0 (1.79) | -0.3 (4.07)
  Change from Baseline - Day 2/36 Hour | 2.0 (4.00) | 6.0 (0) | -1.3 (3.06) | -0.7 (6.43) | -1.0 (3.74) | 0.7 (2.07) | -0.7 (2.07) | -2.0 (3.58) | 0.3 (2.66) | 0.7 (2.42) | 1.3 (3.06) | 0 (2.53) | 0.9 (3.63)
  Change from Baseline - Day 3/42 Hour | -0.7 (3.06) | 3.3 (2.31) | -4.7 (2.31) | 0.7 (6.11) | -0.7 (2.42) | 0.3 (3.44) | 2.7 (3.50) | -1.0 (2.10) | -1.0 (3.29) | 2.0 (1.79) | 1.3 (4.16) | 0.3 (1.97) | 2.9 (2.79)
  Change from Baseline - Day 3/48 Hour | -2.7 (1.15) | 1.3 (2.31) | -0.7 (1.15) | 1.3 (3.06) | -1.7 (4.27) | -0.3 (2.34) | 0.7 (2.07) | 0.3 (2.34) | -0.7 (2.42) | -0.7 (1.63) | -1.3 (3.06) | -0.7 (2.73) | 0.6 (3.95)
  Change from Baseline - Day 4 | -0.7 (6.11) | 4.7 (3.06) | -2.0 (2.00) | 0.7 (3.06) | -1.0 (2.10) | -0.3 (2.34) | 4.0 (1.79) | 1.0 (2.76) | 1.0 (2.76) | 2.3 (3.67) | 0 (5.29) | -0.3 (1.97) | 0.3 (3.15)
  Change from Baseline - Day 7: number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6 | 5 | 6 | 3 | 6 | 7
  Change from Baseline - Day 7 | 1.3 (4.16) | 2.0 (0) | -1.3 (1.15) | 1.3 (5.03) | -2.7 (3.50) | 0.7 (3.01) | 2.7 (3.01) | -1.3 (1.63) | 0.4 (2.61) | 3.7 (1.51) | -0.7 (4.62) | -1.0 (2.10) | 1.7 (2.93)
  Change from Baseline - Day 28 | 0.7 (1.15) | 4.0 (0) | -1.3 (1.15) | 1.3 (3.06) | -2.0 (2.19) | -2.0 (1.26) | 0 (2.19) | -0.7 (2.42) | -0.7 (4.84) | 0.7 (3.27) | 0.7 (4.16) | -0.3 (3.88) | 0.3 (2.69)

7. Primary Outcome: Change In Heart Rate
Description: Heart rate measurements were measured at specific time points.
Time Frame: Days 1, 2, 3, 4, 7 and 28
Population: Safety population: all participants who received any amount of study drug.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Cohort 1: 100 mg PB2452 (no Ticagrelor) | Cohort 2: 300 mg PB2452 (no Ticagrelor) | Cohort 3: 1000 mg PB2452 (no Ticagrelor) | Cohort 1 to 3: Placebo | Cohort 4: 1000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 5: 3000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 6: 9000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 4 to 6: Placebo | Cohort 7: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 8: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 9: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 10: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 7 to 10: Placebo
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 3 | 6 | 7
Beats per minute
  Change from Baseline - Day 1/0.5 Hour: number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6 | 4 | 4 | 3 | 6 | 7
  Change from Baseline - Day 1/0.5 Hour | -8.3 (3.21) | 4.0 (3.46) | -7.0 (6.08) | 3.0 (8.00) | 3.5 (8.12) | -5.5 (3.39) | -0.2 (6.21) | -3.0 (9.53) | -2.5 (5.07) | -5.5 (5.80) | -4.0 (9.54) | -1.0 (3.35) | -4.6 (7.23)
  Change from Baseline - Day 1/0.75 Hour | -3.0 (1.73) | 5.7 (1.53) | -6.7 (4.16) | 5.7 (7.51) | 2.2 (9.06) | -0.2 (5.95) | -5.2 (2.14) | -1.7 (11.64) | 1.5 (3.83) | -5.3 (3.39) | -5.3 (6.66) | 1.3 (5.54) | -2.6 (5.38)
  Change from Baseline - Day 1/1 Hour | -0.3 (1.53) | 4.3 (1.53) | -7.0 (4.58) | 5.7 (9.29) | 2.3 (5.47) | 0 (3.58) | -4.7 (3.88) | -2.0 (10.71) | 0.2 (3.43) | -5.7 (5.13) | -7.3 (7.51) | 1.0 (2.37) | -2.7 (3.59)
  Change from Baseline - Day 1/2 Hour: number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 3 | 5 | 7
  Change from Baseline - Day 1/2 Hour | -3.7 (4.62) | 6.0 (1.00) | -7.3 (6.43) | 1.3 (0.58) | 3.0 (4.10) | 1.7 (5.09) | -5.0 (3.79) | -2.5 (9.79) | 2.7 (11.96) | -5.8 (6.62) | -3.7 (9.71) | -3.2 (0.84) | -2.9 (6.36)
  Change from Baseline - Day 1/4 Hour | -0.3 (2.89) | 13.7 (4.04) | -3.7 (3.21) | 5.0 (8.00) | 5.7 (4.63) | 1.8 (3.82) | 1.5 (7.53) | 3.8 (9.79) | 4.8 (2.56) | -0.2 (6.11) | -0.3 (3.06) | 6.0 (3.58) | 1.6 (7.81)
  Change from Baseline - Day 1/8 Hour: number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 5 | 3 | 6 | 7
  Change from Baseline - Day 1/8 Hour | 1.7 (5.03) | 14.7 (0.58) | -5.7 (4.73) | 7.3 (14.47) | 8.0 (8.32) | 5.8 (7.76) | 3.2 (6.15) | 4.3 (15.42) | 6.5 (2.88) | 4.0 (10.65) | 2.7 (1.53) | 8.5 (6.16) | 5.9 (7.47)
  Change from Baseline - Day 2/24 Hour | -2.0 (3.00) | 9.0 (8.19) | -10.7 (4.73) | -0.3 (4.73) | -3.0 (5.40) | 2.0 (3.85) | 0.8 (5.15) | 0.3 (10.65) | 0.8 (3.87) | -4.5 (4.76) | -2.0 (3.00) | 1.3 (6.41) | -2.4 (5.09)
  Change from Baseline - Day 2/30 Hour | 0 (6.08) | 11.7 (3.21) | 0 (3.61) | 4.3 (4.73) | 10.0 (5.22) | 6.8 (7.28) | 3.2 (6.43) | 3.5 (11.15) | 6.8 (6.55) | 6.3 (6.65) | 0 (4.36) | 8.2 (5.88) | 3.4 (5.50)
  Change from Baseline - Day 2/36 Hour: number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 5 | 6 | 6 | 6 | 6 | 3 | 6 | 7
  Change from Baseline - Day 2/36 Hour | 2.3 (8.50) | 12.0 (9.64) | -2.0 (4.00) | 5.0 (8.54) | 9.0 (6.00) | 7.4 (5.86) | 8.8 (6.85) | 3.2 (11.89) | 8.0 (5.10) | 10.0 (8.88) | 3.3 (3.21) | 12.7 (8.73) | 2.3 (7.74)
  Change from Baseline - Day 3/42 Hour | 2.0 (3.00) | 8.3 (4.04) | -3.0 (5.57) | 2.0 (6.08) | 5.2 (8.89) | -2.5 (2.35) | 4.8 (11.07) | -1.8 (9.47) | 2.0 (6.96) | -1.5 (6.66) | 0.7 (5.51) | 1.5 (5.68) | -0.1 (9.15)
  Change from Baseline - Day 3/48 Hour | -1.0 (7.00) | 10.3 (7.02) | -9.3 (5.86) | -3.3 (5.69) | 2.8 (3.19) | 1.7 (5.82) | -0.2 (5.42) | 2.0 (7.77) | 2.0 (2.00) | -2.8 (6.34) | 1.7 (1.15) | 3.8 (4.79) | -1.1 (5.21)
  Change from Baseline - Day 4 | 6.0 (8.89) | 9.0 (7.55) | -8.3 (7.37) | 1.3 (12.50) | 6.7 (9.03) | 5.2 (9.89) | -3.5 (3.73) | 2.5 (7.74) | 5.0 (5.40) | 3.5 (13.03) | 7.7 (7.77) | 3.5 (8.38) | 1.4 (7.96)
  Change from Baseline - Day 7: number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6 | 5 | 6 | 3 | 6 | 7
  Change from Baseline - Day 7 | -4.3 (3.21) | 8.0 (11.36) | -10.7 (8.74) | 0.3 (11.15) | 4.2 (8.61) | 5.8 (10.57) | -5.8 (5.85) | -4.8 (12.67) | 0.8 (3.96) | -4.5 (8.48) | -12.0 (10.39) | 2.3 (7.31) | 1.7 (7.34)
  Change from Baseline - Day 28 | -7.7 (7.77) | 4.0 (6.56) | -8.3 (8.08) | -9.3 (9.07) | -1.7 (5.54) | -4.0 (3.63) | -6.5 (8.73) | -4.8 (6.85) | -1.0 (3.58) | 0.2 (11.36) | -12.0 (16.00) | -4.7 (1.75) | -0.1 (12.06)

8. Primary Outcome: Incidence of Clinically Significant 12-Lead Electrocardiogram (ECG) Findings
Description: Number of participants per cohort with clinically significant ECG findings.
Time Frame: 60 days - Starting up to 28 days prior to dosing
Population: Safety population: all participants who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: 100 mg PB2452 (no Ticagrelor) | Cohort 2: 300 mg PB2452 (no Ticagrelor) | Cohort 3: 1000 mg PB2452 (no Ticagrelor) | Cohort 1 to 3: Placebo | Cohort 4: 1000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 5: 3000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 6: 9000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 4 to 6: Placebo | Cohort 7: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 8: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 9: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 10: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 7 to 10: Placebo
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 3 | 6 | 7
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Incidence of Clinically Significant Cardiac Telemetry Findings
Description: Number of participants per cohort with clinically significant cardiac telemetry findings.
Time Frame: 3 Days - Starting 1 day prior to dosing up to 2 days after dosing
Population: Safety population: all participants who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: 100 mg PB2452 (no Ticagrelor) | Cohort 2: 300 mg PB2452 (no Ticagrelor) | Cohort 3: 1000 mg PB2452 (no Ticagrelor) | Cohort 1 to 3: Placebo | Cohort 4: 1000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 5: 3000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 6: 9000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 4 to 6: Placebo | Cohort 7: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 8: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 9: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 10: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 7 to 10: Placebo
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 3 | 6 | 7
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: Participants Experiencing Anti-drug Antibodies (ADAs)
Description: Incidence of Immunogenicity.
Time Frame: Day -3, Day -1, Day 7, and Day 28
Population: Safety population: all participants who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- All PB2452: All participants in any cohorts who received PB2452.
- All Placebo: All participants in any cohorts who received placebo.
Arm/Group | Cohort 1: 100 mg PB2452 (no Ticagrelor) | Cohort 2: 300 mg PB2452 (no Ticagrelor) | Cohort 3: 1000 mg PB2452 (no Ticagrelor) | Cohort 1 to 3: Placebo | Cohort 4: 1000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 5: 3000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 6: 9000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 4 to 6: Placebo | Cohort 7: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 8: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 9: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 10: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 7 to 10: Placebo | All PB2452 | All Placebo
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 3 | 6 | 7 | 78 | 16
Participants
  Day -3 | NA — Cohorts 1-3 had baseline testing at Day -1 and Cohorts 4-10 had baseline testing at Day -3. | NA — Cohorts 1-3 had baseline testing at Day -1 and Cohorts 4-10 had baseline testing at Day -3. | NA — Cohorts 1-3 had baseline testing at Day -1 and Cohorts 4-10 had baseline testing at Day -3. | NA — Cohorts 1-3 had baseline testing at Day -1 and Cohorts 4-10 had baseline testing at Day -3. | 1 | 2 | 0 | 1 | 2 | 4 | 0 | 5 | 0 | 14 | 1
  Day -1 | 1 | 0 | 0 | 1 | NA — Cohorts 1-3 had baseline testing at Day -1 and Cohorts 4-10 had baseline testing at Day -3. | NA — Cohorts 1-3 had baseline testing at Day -1 and Cohorts 4-10 had baseline testing at Day -3. | NA — Cohorts 1-3 had baseline testing at Day -1 and Cohorts 4-10 had baseline testing at Day -3. | NA — Cohorts 1-3 had baseline testing at Day -1 and Cohorts 4-10 had baseline testing at Day -3. | NA — Cohorts 1-3 had baseline testing at Day -1 and Cohorts 4-10 had baseline testing at Day -3. | NA — Cohorts 1-3 had baseline testing at Day -1 and Cohorts 4-10 had baseline testing at Day -3. | NA — Cohorts 1-3 had baseline testing at Day -1 and Cohorts 4-10 had baseline testing at Day -3. | NA — Cohorts 1-3 had baseline testing at Day -1 and Cohorts 4-10 had baseline testing at Day -3. | NA — Cohorts 1-3 had baseline testing at Day -1 and Cohorts 4-10 had baseline testing at Day -3. | 1 | 1
  Day 7 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 1 | 4 | 0 | 2 | 0 | 11 | 3
  Day 28 | 1 | 0 | 1 | 0 | 2 | 2 | 1 | 1 | 5 | 4 | 0 | 5 | 0 | 21 | 1

11. Primary Outcome: Maximal Percent of Baseline Platelet Aggregation (PA(Max)) in Cohorts 4-6
Description: Effectiveness Of Single Ascending Doses Of PB2452. IPA [maximum (max)] induced by 20 µM adenosine diphosphate (ADP) at each assessment point.
Time Frame: Before dosing and at 0.5, 1, 2, 3, 6, 12, 24, and 48 hours after PB2452 infusion and 5th ticagrelor dose.
Population: Pharmacodynamic (PD) Population: all participants who received at least 1 dose of ticagrelor and had at least 1 measurable post dose light transmission aggregometry (LTA) value.
  PD samples were not collected for participants in Cohorts 1 to 3; therefore, they were not included in the PD Population.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Cohort 4 to 6: Placebo | Cohort 4: 1000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 5: 3000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 6: 9000 mg PB2452 (Ticagrelor Pre-Trx)
Number analyzed (Participants) | 6 | 6 | 6 | 6
percentage | 77.1 (14.5) | 67.9 (18.3) | 92.6 (9.2) | 97.3 (3.9)

12. Primary Outcome: Final Extent Percent of Baseline Platelet Aggregation in Cohorts 4-6
Description: Effectiveness Of Single Ascending Doses Of PB2452. IPA [final extent] induced by 20 µM adenosine diphosphate (ADP) at each assessment point.
Time Frame: Before dosing and at 0.5, 1, 2, 3, 6, 12, 24, and 48 hours after PB2452 infusion and 5th ticagrelor dose.
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Cohort 4 to 6: Placebo | Cohort 4: 1000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 5: 3000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 6: 9000 mg PB2452 (Ticagrelor Pre-Trx)
Number analyzed (Participants) | 6 | 6 | 6 | 6
percentage | 66.5 (30.3) | 58.4 (27.0) | 90.6 (9.7) | 94.6 (9.3)

13. Primary Outcome: Maximal Actual Platelet Aggregation (APA(Max)) (Cohorts 4-6)
Description: Effectiveness Of Single Ascending Doses Of PB2452 - Inhibition of maximal platelet aggregation.
Time Frame: Before dosing and at 0.5, 1, 2, 3, 6, 12, 24, and 48 hours after PB2452 infusion and 5th ticagrelor dose. And at 1, 2, 6, and 12 hours after the Day 2 post-MEDI2452 (PB2452) 6th ticagrelor dose (Cohorts 8 and 9 Only).
Population: PD Population: all participants who received at least 1 dose of ticagrelor and had at least 1 measurable post dose LTA value.
  PD samples were not collected for participants in Cohorts 1 to 3, therefore, they were not included in the PD Population.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Cohort 4 to 6: Placebo | Cohort 4: 1000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 5: 3000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 6: 9000 mg PB2452 (Ticagrelor Pre-Trx)
Number analyzed (Participants) | 6 | 6 | 6 | 6
percentage | 61.7 (13.3) | 59.5 (15.1) | 77.5 (8.4) | 83.7 (13.8)

14. Primary Outcome: Time to Maximum Platelet Aggregation (TPA(Max)) (Cohorts 4-6)
Description: Effectiveness Of Single Ascending Doses Of PB2452 - Time to IPAmax.
Time Frame: Before dosing and at 0.5, 1, 2, 3, 6, 12, 24, and 48 hours after PB2452 infusion and 5th ticagrelor dose.
Population: as for outcome 13
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 4 to 6: Placebo | Cohort 4: 1000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 5: 3000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 6: 9000 mg PB2452 (Ticagrelor Pre-Trx)
Number analyzed (Participants) | 6 | 6 | 6 | 6
hours | 48.00 [48.00 to 48.00] | 48.00 [48.00 to 48.10] | 0.51 [0.50 to 1.00] | 0.82 [0.50 to 2.12]

15. Primary Outcome: Maximal Percent of Baseline Platelet Aggregation (PA(Max)) (Cohorts 7-10)
Description: Effectiveness Of Single Ascending Doses Of PB2452 - IPA (max) induced by 20 µM ADP at each assessment point.
Time Frame: Before dosing and at 5 min, 0.25, 0.5, 1, 2, 3, 6, 8, 10, 12, 16, 20, 24, and 48 hours after PB2452 infusion and 5th ticagrelor dose. And at 1, 2, 6, and 12 hours after the Day 2 post-MEDI2452 (PB2452) 6th ticagrelor dose.
Population: PD Population: all participants who received at least 1 dose of ticagrelor and had at least 1 measurable post dose LTA value.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Cohort 7 to 10: Placebo | Cohort 7: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 8: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 9: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 10: 18000 mg PB2452 (Ticagrelor Pre-Trx)
Number analyzed (Participants) | 7 | 6 | 6 | 3 | 6
percentage | 62.2 (20.1) | 98.9 (2.8) | 98.6 (3.0) | 100.0 (0) | 98.7 (2.1)

16. Primary Outcome: Final Extent Percent of Baseline Platelet Aggregation (Cohorts 7-10)
Description: Effectiveness Of Single Ascending Doses Of PB2452 - IPA (max) induced by 20 µM ADP at each assessment point.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Cohort 7 to 10: Placebo | Cohort 7: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 8: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 9: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 10: 18000 mg PB2452 (Ticagrelor Pre-Trx)
Number analyzed (Participants) | 7 | 6 | 6 | 3 | 6
percentage | 51.5 (26.4) | 96.1 (9.6) | 98.2 (3.4) | 100.0 (0) | 97.3 (4.7)

17. Primary Outcome: Maximal Actual Platelet Aggregation (APA(Max)) (Cohorts 7-10)
Description: Effectiveness Of Single Ascending Doses Of PB2452 - Inhibition of maximal platelet aggregation.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Cohort 7 to 10: Placebo | Cohort 7: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 8: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 9: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 10: 18000 mg PB2452 (Ticagrelor Pre-Trx)
Number analyzed (Participants) | 7 | 6 | 6 | 3 | 6
percentage | 51.9 (17.8) | 84.8 (9.3) | 86.0 (5.7) | 94.7 (1.2) | 86.0 (2.8)

18. Primary Outcome: Time to Maximum Platelet Aggregation (TPA(Max))(Cohorts 7-10)
Description: Effectiveness Of Single Ascending Doses Of PB2452 - Time to IPAmax
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 7 to 10: Placebo | Cohort 7: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 8: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 9: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 10: 18000 mg PB2452 (Ticagrelor Pre-Trx)
Number analyzed (Participants) | 7 | 6 | 6 | 3 | 6
hours | 48.00 [3.00 to 48.05] | 6.00 [2.00 to 16.00] | 5.50 [0.53 to 16.00] | 6.00 [1.02 to 8.00] | 1.25 [0.25 to 48.00]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from Day -3 (Cohorts 4 through 10) or Day -1 (Cohorts 1 through 3) until completion of all study procedures and EOS assessments (Day 28).
Arm/Group | Cohort 1: 100 mg PB2452 (no Ticagrelor) | Cohort 2: 300 mg PB2452 (no Ticagrelor) | Cohort 3: 1000 mg PB2452 (no Ticagrelor) | Cohort 1 to 3: Placebo | Cohort 4: 1000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 5: 3000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 6: 9000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 4 to 6: Placebo | Cohort 7: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 8: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 9: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 10: 18000 mg PB2452 (Ticagrelor Pre-Trx) | Cohort 7 to 10: Placebo | All PB2452 | All Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/3 | 0/6 | 0/7 | 0/48 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 1/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/3 | 0/6 | 0/7 | 1/48 | 0/16
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 1/3 | 1/3 | 3/6 | 0/6 | 6/6 | 1/6 | 2/6 | 2/6 | 1/3 | 2/6 | 0/7 | 17/48 | 2/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: 100 mg PB2452 (no Ticagrelor) (N=3) | Cohort 2: 300 mg PB2452 (no Ticagrelor) (N=3) | Cohort 3: 1000 mg PB2452 (no Ticagrelor) (N=3) | Cohort 1 to 3: Placebo (N=3) | Cohort 4: 1000 mg PB2452 (Ticagrelor Pre-Trx) (N=6) | Cohort 5: 3000 mg PB2452 (Ticagrelor Pre-Trx) (N=6) | Cohort 6: 9000 mg PB2452 (Ticagrelor Pre-Trx) (N=6) | Cohort 4 to 6: Placebo (N=6) | Cohort 7: 18000 mg PB2452 (Ticagrelor Pre-Trx) (N=6) | Cohort 8: 18000 mg PB2452 (Ticagrelor Pre-Trx) (N=6) | Cohort 9: 18000 mg PB2452 (Ticagrelor Pre-Trx) (N=3) | Cohort 10: 18000 mg PB2452 (Ticagrelor Pre-Trx) (N=6) | Cohort 7 to 10: Placebo (N=7) | All PB2452 (N=48) | All Placebo (N=16)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: 100 mg PB2452 (no Ticagrelor) (N=3) | Cohort 2: 300 mg PB2452 (no Ticagrelor) (N=3) | Cohort 3: 1000 mg PB2452 (no Ticagrelor) (N=3) | Cohort 1 to 3: Placebo (N=3) | Cohort 4: 1000 mg PB2452 (Ticagrelor Pre-Trx) (N=6) | Cohort 5: 3000 mg PB2452 (Ticagrelor Pre-Trx) (N=6) | Cohort 6: 9000 mg PB2452 (Ticagrelor Pre-Trx) (N=6) | Cohort 4 to 6: Placebo (N=6) | Cohort 7: 18000 mg PB2452 (Ticagrelor Pre-Trx) (N=6) | Cohort 8: 18000 mg PB2452 (Ticagrelor Pre-Trx) (N=6) | Cohort 9: 18000 mg PB2452 (Ticagrelor Pre-Trx) (N=3) | Cohort 10: 18000 mg PB2452 (Ticagrelor Pre-Trx) (N=6) | Cohort 7 to 10: Placebo (N=7) | All PB2452 (N=48) | All Placebo (N=16)
Infusion site bruising (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 0
Medical device site reaction (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Vessel puncture site bruise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0
Infusion site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aspiration Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eyelid irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Blood urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT03492385/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-12): https://cdn.clinicaltrials.gov/large-docs/85/NCT03492385/SAP_001.pdf